CLINICAL TRIAL: NCT00793130
Title: The Efficacy and Tolerability of Coltect as Add-on in Patients With Active Ulcerative Colitis - an Open Label
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Iris Dotan, Department of Gastroenterology and Liver Diseases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-08-ID-348-CTIL
Record Dates: First submitted 2008-11-16; First posted 2008-11-19 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative; Colitis; Coltect; Curcumin; Green tea; Selenium; inflammation; bowel
MeSH Terms: conditions — Colitis, Ulcerative; Ulcer; Colitis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Coltect (Other): Coltect contains natural compounds: curcumin, green tea and selenium which are approved as food supplements by the Ministry of Health in Israel. Curcumin and green tea are widely used in the food industry.
  Interventions: Dietary Supplement: Coltect

INTERVENTIONS:
Dietary Supplement: Coltect — Two tablets twice daily (BID) during the 2 months of the study. Each tablet contains 500mg Curcumin, 250mg Green tea and 100mcg Selenomethionine.

SUMMARY:
The aim of the study is to reduce the severity and duration of acute attacks, to prevent the recurrence of new acute attacks and to improve patient's quality of life.

Coltect contains anti inflammatory and antioxidant natural agents (curcumin, green tea and selenomethionine) which are associated with a positive effect on inflammatory disease.

The investigators assume that Coltect represents a tolerable and mild treatment, viable alternative to other medical therapies with fewer side effects.

Coltect is a food supplement that contains active ingredients from herbal sources.

DETAILED DESCRIPTION:
Studies in animal models of colitis and in humans with IBD demonstrated that the components of Coltect have anti-inflammatory effects:

Hanai H. et al demonstrated that curcumin was safe and effective in maintaining remission in patients with quiescent UC. (7)

B.Salh et al showed that curcumin, was able to attenuate colitis in the dinitrobenzene sulfonic acid (DNB)-induced murine model of colitis. The immunohistochemical signal is dramatically attenuated at the level of the mucosa by curcumin. The authors thus proposed that curcumin may have therapeutic implications for human IBD. (8)

Potential Benefits of Coltect- Coltect might be suited for the treatment of patients with mild to moderate flare-ups of ulcerative colitis.

Coltect provides an effect with expected low incidence of side effects. (each agent tested before and found safe for human use).

The availability of a safe and effective non-surgical and non steroids treatment of active ulcerative colitis.

Overview - Clinical indication and summary of existing preclinical and clinical knowledge pertaining to the product.

Coltect contains natural compounds: curcumin, green tea and selenium which are approved as food supplements by the Ministry of Health in Israel. Curcumin and green tea are widely used in the food industry.

Curcumin is a natural compound found in the plant Curcuma longa which is used as a food additive known as turmeric. The major pigment in turmeric is curcumin - chemical name diferuloymethane, which possesses both anti-inflammatory and antioxidant properties. Curcumin also strongly inhibits proliferation of HT-29 and HCT-15 human colon cancer cell lines (1). Dietary administration of curcumin suppresses the development of chemically induced cancers(1). These properties have led to studies on the chemopreventive effects of curcumin which also showed that the agent reduces colonic inflammatory responses.

Curcumin has a profound immunosuppressive effect via inhibition of IL-2 synthesis as well as IL-2 and mitogen activation of human leukocytes. This immunosuppressive effect may be mediated by NFκB inhibition (1).

Based on the aforementioned, curcumin appears to reduce the inflammatory response in ulcerative colitis patients Clinical studies with curcumin have shown beneficial effects in experimental studies of acute and chronic diseases characterized by an exaggerated inflammatory reaction. There is an ample evidence to support its clinical use both in the prevention and a treatment setting. Several natural substances such as curcumin have greater antioxidant effects than conventional vitamins, including various polyphenols, flavonoids and curcumenoids. Natural substances are worth further research both experimentally and clinically.

Sting et al found that: Curcumin was shown to be non-toxic, to have antioxidant activity, and to inhibit such mediators of inflammation such as NFkB, cyclooxygenase-2 (COX-2), lipooxygenase (LOX), and inducible nitric oxide synthase (iNOS). (13)

Ricky A. Sharma et al designed a dose-escalation study to explore the pharmacology of curcumin in humans. Patients with advanced colorectal cancer consumed capsules compatible with curcumin doses between 0.45 and 3.6gr. daily for up to 4 months. Curcumin was well tolerated at all of the dose levels, and dose-limiting toxicity was not observed. At dose of 3.6gr. mild diarrhea is only discernible toxicity. (2) Cheng et al. treated patients with pre-malignant conditions with tablets containing pure curcumin for up to 3 months at daily dose as high as 8gr. without evident toxicity . They recommended that the common therapeutic dose would be 400-600 mg curcumin 3 times daily.(14)

Ricky el al showed that consumption of 3.6 g of curcumin daily causes inhibition of PGE2 production by blood leukocytes measured ex vivo.(2)

In therapy for UC, a double blind placebo-controlled trial with curcumin found that both the clinical and endoscopic evaluation scores were significantly improved by curcumin therapy. The endoscopic score was substantially improved compared with the placebo.

The results of this study indicate that the turmeric component, curcumin, is potentially a promising medication for the treatment of IBD (7)

Green tea is made from unfermented, solely leaves of Camellia sinensis and contains the highest concentration of powerful antioxidants called polyphenols.

The green tea polyphenols include (-)-epigallocatechin gallate (EGCG), (-) epigallocatechin (EGC), (-)-epicatechin gallate (ECG) and (-)-epicatechin (EC), they have potent antioxidant properties. (9) Gary et al provide evidence that green tea polyphenols have anti-inflammatory effects in murine colitis. They showed that mice treated with green tea polyphenols have less severe colitis, and green tea polyphenols are widely distributed throughout the body, one of the highest tissue concentrations is found in the intestine. This distribution favors its use in gastrointestinal diseases such as IBD.(9)

Selenium is an essential trace element with a worldwide average nutritional intake of 50 to 350 µg/d function as an antioxidant and anti inflammatory and associated with colorectal cancer prevention.(10,11) Marwan et al established the safety of administering high dose (2200 µg) of selenomethionine in humans with cancer up to 13 months. (12) Toxicity at high dose selenium appeared as mild headache, nausea or heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old.
* Subjects with mild to moderate active ulcerative colitis
* Hemoglobin value greater than 10 g/dL.
* Aspartate aminotransferase and alanine aminotransferase <1.5 times the upper limit of normal.
* Serum bilirubin and creatinine <1.5 × upper limit of normal.
* Subjects that provided informed consent and agree to comply with all study procedure.
* Subjects had a Clinical Activity Index (CAI) >4
* Subjects had a Clinical Activity Index (CAI) ≤8
* Established or new diagnosis.
* Subjects that agreed to undergo sigmoidoscopy at study completion

Exclusion Criteria:

* Active chronic inflammatory or autoimmune disease other than UC.
* Active infection, including viral infection.
* Active peptic ulcer disease.
* Infectious/ Ischemic colitis.
* Acute or chronic cardiac, renal failure (serum creatinine >300 mmol/L)
* Abnormal liver function - (liver function tests greater than 1.5 times upper range of normal).
* Crohn's disease.
* Use of rectal corticosteroids within 4 weeks before study entry.
* Patients with known or suspected bleeding tendency.
* Patients with severe active ulcerative colitis.
* Present or a history of colorectal cancer.
* Serious other disease(s) that according to physicians judgment should preclude the patient from participation in the study.
* Toxic megacolon.
* Prior bowel resection.
* Baseline positive stool culture or C DIFF toxin assay.
* Existing or intended pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
50% improvement of the Clinical Activity Index (CAI) of the study. | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Gush-Dan, Israel